CLINICAL TRIAL: NCT04711213
Title: A Phase 2 Clinical Study to Assess the Efficacy and Safety of SED80 for the Treatment of Inflammation and Pain Associated With Cataract Surgery
Brief Title: A Clinical Study to Assess the Efficacy and Safety of SED80 for Use in Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: iDrop, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-02
Record Dates: First submitted 2020-09-23; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-09

CONDITIONS: Cataract in Inflammatory Ocular Disorders

STUDY DESIGN:
Intervention Model Description: Randomized to 2 active dosing groups and 2 corresponding dosing groups
Who Masked: Participant
Masking Description: Single Masked randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dexamethasone Dose 1 (Active Comparator)
  Interventions: Drug: Dexamethasone Dose 1
- Dexamethasone Dose 2 (Active Comparator)
  Interventions: Drug: Dexamethasone Dose 2
- Placebo Dose 1 (Placebo Comparator)
  Interventions: Drug: Placebo Dose 1
- Placebo Dose 2 (Placebo Comparator)
  Interventions: Drug: Placebo Dose 2

INTERVENTIONS:
Drug: Dexamethasone Dose 1 — Dexamethasone ophthalmic suspension dose 1
  Arms: Dexamethasone Dose 1
Drug: Dexamethasone Dose 2 — Dexamethasone ophthalmic suspension dose 2
  Arms: Dexamethasone Dose 2
Drug: Placebo Dose 1 — Placebo suspension dose 1
  Arms: Placebo Dose 1
Drug: Placebo Dose 2 — Placebo suspension dose 2
  Arms: Placebo Dose 2

SUMMARY:
Patients at least 40 years of age who are undergoing cataract surgery will be randomized to receive treatment with one of four groups of dexamethasone ophthalmic suspension or placebo eye drops to determine if the drops decrease inflammation and pain inside the eye and are safe after cataract surgery.

DETAILED DESCRIPTION:
"Patients undergoing traditional cataract surgery routinely develop inflammation and pain. This study will evaluate 4 arms of either dexamethasone or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing traditional cataract surgery.

Exclusion Criteria:

* Patients with unusual ocular conditions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Ocular inflammation | Day 8
  Measuring Anterior Cell Count

SECONDARY OUTCOMES:
Ocular Pain | Day 8
  Measuring patient ocular pain using an 11-point visual scale

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Casada, MD, Principal Investigator — President - Centre De. Oftalmolgia
Locations (1):
- Centre De. Oftalmologia, San Salvador, El Salvador

IPD SHARING:
Plan to Share IPD: No